CLINICAL TRIAL: NCT06843460
Title: A Single-Dose Clinical Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Sotatercept (MK-7962) in Healthy Chinese Participants
Brief Title: A Clinical Study of MK-7962 in Healthy Chinese Participants (MK-7962-021)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 7962-021
Record Dates: First submitted 2025-02-20; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Healthy
MeSH Terms: interventions — ACE-011

STUDY DESIGN:
Intervention Model Description: The first 12 participants were randomized 1:3 between placebo or 0.3 mg/kg of sotatercept. After those 12 participants were complete, the next 12 were randomized 1:3 between placebo or 0.7 mg/kg of sotatercept.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Sotatercept Dose Level 1 (Experimental): Participants received a single dose of sotatercept at dose level 1.
  Interventions: Biological: Sotatercept
- Sotatercept Dose Level 2 (Experimental): Participants received a single dose of sotatercept at dose level 2.
  Interventions: Biological: Sotatercept
- Placebo (Placebo Comparator): Participants received a single dose of placebo to sotatercept.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Sotatercept — Single subcutaneous injection
  Other Names: MK-7962; ActRIIA-IgG1Fc; ACE-011
  Arms: Sotatercept Dose Level 1; Sotatercept Dose Level 2
Other: Placebo — Single subcutaneous injection
  Arms: Placebo

SUMMARY:
The goal of this study is to learn about the safety of 2 different amounts of sotatercept and if healthy Chinese people tolerate them. The study will also measure what happens to sotatercept in a person's body over time (pharmacokinetic or PK study).

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Is in good health
* Has a BMI≥18.0 kg/m^2 and ≤28.0 kg/m^2

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* Has a history of clinically significant endocrine, GI, cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, or major neurological (including stroke and chronic seizures) abnormalities or diseases
* Has been treated with a sotatercept or luspatercept

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2023-11-22 (Actual); Primary Completion 2024-05-21 (Actual); Study Completion 2024-05-21 (Actual)

PRIMARY OUTCOMES:
Number of Participants Who Experience an Adverse Event (AE) | Up to approximately 120 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who experience an AE will be reported.
Number of Participants Who Discontinue Study Due to an AE | Up to approximately 120 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who discontinue study due to an AE will be reported.
Maximum Serum Concentration (Cmax) of Sotatercept | At designated timepoints (up to 120 days)
  Blood samples will be collected to determine the Cmax of sotatercept.
Time to Maximum Serum Concentration (Tmax) of Sotatercept | Predose and at designated timepoints up to 120 days postdose
  Blood samples will be collected to determine the Tmax of sotatercept.
Area Under the Concentration-Time Curve from Time 0 to Last (AUC0-Last) of MK-7962 | At designated timepoints (up to 120 days)
  Blood samples will be collected to determine the AUC0-last of MK-7962.
Area Under the Concentration-Time Curve from Time 0 to Infinity (AUC0-Inf) of MK-7962 | At designated timepoints (up to 120 days)
  Blood samples will be collected to determine the AUC0-inf of MK-7962.
Area Under the Concentration-Time Curve from Time 0 to 28 days (AUC0-28 days) of MK-7962 | At designated timepoints (up to 28 days postdose)
  Blood samples will be collected to determine the AUC0-28 days of MK-7962.
Apparent Terminal Half-life (t1/2) of MK-7962 | At designated timepoints (up to 120 days)
  Blood samples will be collected to determine the t1/2 of MK-7962.
Apparent Clearance (CL/F) of MK-7962 | At designated timepoints (up to 120 days)
  Blood samples will be collected to determine the CL/F of MK-7962.
Apparent Volume of Distribution During Terminal Phase (Vz/F) of MK-7962 | At designated timepoints (up to 120 days)
  Blood samples will be collected to determine the Vz/F of MK-7962.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Zhongshan Hospital,Fudan University-Dep. of Clinical Pharmacology (Site 0001), Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com